CLINICAL TRIAL: NCT01121276
Title: A Trial Investigating the Pharmacodynamic Properties of NN1218 in Subjects With Type 1 and Type 2 Diabetes
Brief Title: A Trial Investigating NN1218 in Subjects With Type 1 and Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN1218-3824; U1111-1113-6897 (Other: WHO); 2009-017627-25 (EudraCT Number)
Record Dates: First submitted 2010-05-10; First posted 2010-05-12 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — Insulin Aspart

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- NN1218, formulation A (Experimental)
  Interventions: Drug: Faster-acting insulin aspart
- NN1218, formulation B (Experimental)
  Interventions: Drug: Faster-acting insulin aspart
- NN1218, formulation C (Experimental)
  Interventions: Drug: Faster-acting insulin aspart
- NN1218, formulation D (Experimental)
  Interventions: Drug: Faster-acting insulin aspart
- insulin aspart (Active Comparator)
  Interventions: Drug: insulin aspart

INTERVENTIONS:
Drug: Faster-acting insulin aspart — 0.2 U/kg body weight injected subcutaneously (under the skin)
  Other Names: NN1218
  Arms: NN1218, formulation A
Drug: insulin aspart — 0.2 U/kg body weight injected subcutaneously (under the skin)
  Arms: insulin aspart
Drug: Faster-acting insulin aspart — 0.2 U/kg body weight injected subcutaneously (under the skin)
  Other Names: NN1218
  Arms: NN1218, formulation B
Drug: Faster-acting insulin aspart — 0.2 U/kg body weight injected subcutaneously (under the skin)
  Other Names: NN1218
  Arms: NN1218, formulation C
Drug: Faster-acting insulin aspart — 0.2 U/kg body weight injected subcutaneously (under the skin)
  Other Names: NN1218
  Arms: NN1218, formulation D

SUMMARY:
This trial is conducted in Europe and in the United States of America (USA). The aim of this trial is to investigate the absorption and effect in the body of NN1218 in subjects with type 1 and type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or type 2 diabetes mellitus for more than 12 months
* Treated with multiple daily insulin injections or continuous subcutaneous insulin infusion (CSII) for 12 months or longer for subjects with type 1 diabetes and for 3 months or longer for subjects with type 2 diabetes
* Body Mass Index (BMI) between 18.0-32.0 kg/m2 (both inclusive)

Exclusion Criteria:

* Surgery or trauma with significant blood loss (more than 500 mL) within the last 3 months prior to trial start
* Smoker (defined as a subject who is smoking more than 5 cigarettes or the equivalent per day)
* Not able or willing to refrain from smoking and use of nicotine gum or transdermal nicotine patches during the inpatient period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2010-04; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Area under the blood glucose concentration-time curve | from 0-2 hours

SECONDARY OUTCOMES:
Area under the blood glucose concentration-time curve | from 0-6 hours

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Chula Vista, California, United States

REFERENCES:
- [Background] Heise T, Haahr H, Jensen L, Ericsen L, Hompesch M. Faster-acting Insulin Aspart Improves Postprandial Glycemia vs Insulin Aspart in Patients with Type 1 Diabetes Mellitus (T1DM). Diabetes 2014; 63 ((Suppl 1)): A34 (abstract 129-OR)
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com